CLINICAL TRIAL: NCT07362693
Title: A Prospective, Multicenter, Observational Cohort Study on the Efficacy and Safety of Biological Agents in Patients With Allergic Bronchopulmonary Aspergillosis
Brief Title: A Cohort Study of the Efficacy and Safety of Biologics in Patients With ABPA
Status: Not yet recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Prof., Qianfoshan Hospital
Other Study IDs: ABPA-002
Record Dates: First submitted 2025-12-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: ABPA; Biologics; Allergic Bronchopulmonary Aspergillosis (ABPA); Cohort Study; Allergic Bronchopulmonary Aspergillosis; Efficacy and Safety
Keywords: abpa; Allergic Bronchopulmonary Aspergillosis; Biologics
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary; Invasive Pulmonary Aspergillosis | interventions — Biological Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum, plasma, sputum, bronchoalveolar lavage fluid, stool, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observation group: on the basis of the original standard drug treatment, combined with biological ag
  Interventions: Drug: Biologic Agent
- The control group only received standard drug treatment (oral glucocorticoids with or without oral a: The standard medical regimen was oral prednisone (0.5mg/Kg/ day for 4 weeks, 0.25mg/Kg/ day for 4 weeks, followed by 0.125mg/Kg/ day for 4 weeks, followed by a reduction of 5mg every 2 weeks until discontinuation) with or without oral voriconazole (200mg bid, 1 hour before or after meals).

INTERVENTIONS:
Drug: Biologic Agent — On the basis of the original standard drug treatment, biological agents were combined. All patients received at least 4 months of the same biologic agent, as recommended by the GINA2025 guidelines and assessed for response. It can be administered simultaneously with standard medical therapy or as maintenance therapy for 4 months on standard medical therapy. The previous treatment for bronchial asthma was maintained, including inhaled corticosteroids + long-acting β-receptor agonists, leukotriene receptor antagonists, etc.
  Groups: Observation group: on the basis of the original standard drug treatment, combined with biological ag

SUMMARY:
To evaluate the efficacy and safety of biological agents in patients with allergic bronchopulmonary aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of allergic bronchopulmonary aspergillosis, according to the ISHAM guidelines for the diagnosis and treatment of allergic bronchopulmonary aspergillosis (2024 revision).
2. The underlying disease was bronchial asthma, and it was severe bronchial asthma.
3. Have had an acute asthma attack in the past year. Acute exacerbation of asthma is defined as the sudden onset of wheezing, shortness of breath, cough, chest tightness and other symptoms beyond the definition of uncontrolled asthma, or the aggravation of the original symptoms, and is characterized by decreased expiratory flow, often induced by exposure to allergens, irritants or respiratory tract infection.
4. Blood eosinophil count ≥150 cells /μL.
5. Age ≥ 18 years old.

Exclusion Criteria:

1. The underlying diseases were chronic obstructive pulmonary disease and bronchiectasis;
2. Known allergic history to biological agents;
3. Human immunodeficiency virus infection, active pulmonary tuberculosis or pulmonary malignant tumor;
4. Complicated with other diseases requiring long-term systemic use of glucocorticoids or immunosuppressants (such as autoimmune diseases);
5. Pregnant or lactating women;
6. Currently participating in other interventional clinical research;
7. Any other conditions considered by the investigator to preclude participation in the study (e.g., nonadherence, predicted survival <1 year, or severe mental illness that prevented cooperation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with allergic bronchopulmonary aspergillosis included patients with newly diagnosed allergic bronchopulmonary aspergillosis and severe asthma, patients with refractory allergic bronchopulmonary aspergillosis, and patients with treatment-dependent allergic bronchopulmonary aspergillosis.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations (annual exacerbation rate) | 1 year and 2years
  Acute exacerbations include acute exacerbation of allergic bronchopulmonary aspergillosis, acute exacerbation/attack of asthma, and acute exacerbation/bronchiectasis of infection.
  Acute exacerbation of allergic bronchopulmonary aspergillosis: in patients who have been diagnosed with allergic bronchopulmonary aspergillosis, persistent (>14 days) clinical deterioration or worsening of imaging findings, accompanied by an increase in total serum IgE of >50% from the last recorded value in the stable period, with no other cause of deterioration.
  Acute asthma exacerbation/exacerbation: worsening of respiratory symptoms for at least 48 hours without evidence of immunological or radiographic worsening of allergic bronchopulmonary aspergillosis; Acute exacerbation of infectious/bronchiectasis: clinical worsening for at least 48 hours, including cough, dyspnea, changes in sputum volume or texture, sputum purulence, fatigue, malaising, fever, or hemoptysis, without immunological or imaging worse

SECONDARY OUTCOMES:
8-week treatment response rate | 8 weeks
Number of hospitalizations due to acute exacerbations of allergic bronchopulmonary aspergillosis | 2 years
The time to the first exacerbation | 2 years
The number of times achieved remission | 2 years
Daily oral glucocorticoid use rate/average daily oral glucocorticoid dose/cumulative oral glucocorticoid dose | 2 years
Proportion of patients who remain in remission after glucocorticoids are stopped | 2 years
The use of antifungal drugs | 2 years
asthma control test(ACT) | 2 years
Serum total IgE | 2 years
All-cause mortality | 2 years
Aspergillus fumigatus sIgE | 2 years
Aspergillus fumigatus sIgG | 2 years
peripheral blood eosinophil count | 2 years
Results of exhaled nitric oxide test | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, #16766, Jingshi Road, Jinan City, Shandong Province, China, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No